CLINICAL TRIAL: NCT04879797
Title: Reducing Racial Disparities in SMM: Assessing the Integration of Maternal Safety Bundles and Community Based Doulas to Improve Outcomes for Black Women
Brief Title: Reducing Racial Disparities in Severe Maternal Morbidity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tufts University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Baystate Medical Center (Other); Beth Israel Medical Center (Other); Boston Medical Center (Other); UMass Memorial Health (Other); Steward St. Elizabeth's Medical Center of Boston, Inc. (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ndidiamaka Amutah-Onukagha, Associate Professor, Tufts University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M530001 NIH172; 1R01MD016026-01 (NIH)
Record Dates: First submitted 2021-03-17; First posted 2021-05-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Maternal Death
MeSH Terms: conditions — Maternal Death

STUDY DESIGN:
Intervention Model Description: Hybrid type 1 implementation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Safety Bundles Implementation (Other): The first intervention targets obstetric hemorrhage, severe hypertension and maternal health equity by implementing three relevant AIM bundles: Obstetric Hemorrhage, Severe Hypertension in Pregnancy, and Reduction of Peripartum Racial/Ethnic Disparities. The Perinatal Neonatal Quality Improvement Network (PNQIN) will facilitate this collaborative QI project and support participating hospitals by providing guidance, education, and technical assistance to hospitals to support implementation of bundles using the QI process. Implementation strategies are based on the Institute for Healthcare Improvement (IHI) improvement model and the AIM program implementation toolkit and have previously been used by PNQIN to implement the Obstetric Care for Women with Opioid Use Disorder AIM bundle in 22 hospitals, including the five hospitals for this study.
  Interventions: Other: Implementation of Maternal Safety Bundles
- Doula Services (Other): The second intervention that this study evaluates is doula services. Investigators are evaluating doula services that are offered by two doula organizations at three hospitals. Investigators will provide top-up training to these doulas in order to provide some standardization and quality assurance of the services delivered. The training is developed and delivered by an obstetrician (Meadows) and doula (Gebel) and will take place among providers (staff associated with three chosen hospitals), patient navigators, and two doula groups, Birth Sisters and Accompany Doula Care, on factors that comprise the risk profile and how to offer targeted doula services to women who fit the risk profile. All sites will use standardized data instruments to evaluate the number of factors in the risk profile being met as well as standardized language and recruitment materials for mothers.
  Interventions: Other: Doula Services

INTERVENTIONS:
Other: Implementation of Maternal Safety Bundles — In the second phase, implementation of the bundles will take place. During this phase investigators will conduct quarterly surveys with the health facilities to measure implementation progress, including an index of evidence-based practices. Investigators will conduct surveys with postpartum women to measure their patient experience. Surveys will be conducted using RedCap software. Participants will be given the opportunity to complete the survey online or if they prefer, a research assistant can call them to conduct the survey over the phone. Data on SMM will be collected through PELL
  Arms: Maternal Safety Bundles Implementation
Other: Doula Services — Investigators are evaluating doula services that are offered by two doula organizations at three hospitals.
  Arms: Doula Services

SUMMARY:
There is a paucity of research examining the intersection of race, ethnicity, maternal safety bundles, doulas, and maternal outcomes in Black women at increased risk of severe maternal morbidity and mortality. The proposed mixed-methods study is the first systematic investigation of pregnancy complications and outcomes among Black women with whom maternal safety bundles are being implemented including racial disparities, hemorrhage, and hypertension. Additionally, through the analysis of secondary state level data, this study will examine perinatal care, maternal outcomes, and healthcare utilization of Black women at increased risk of severe maternal morbidity and mortality compared with non-Latino white women. Finally, through individual interviews with Black women and focus groups with obstetric health providers and doulas, the study will examine disparities and improve care by creating and disseminating a set of practice recommendations for maternity care for Black women at increased risk of morbidity and mortality.

Research has not yet examined the intersection of race/ethnicity, doulas, and quality improvement (QI) interventions, such as maternal safety bundles, on reducing SMM and mortality among non-Hispanic Black (NHB) women. The overall goal of this mixed-methods study is to use analysis of existing big data and the evaluation of two interventions to ultimately develop targeted recommendations for addressing these inequities. Our approach leverages multiple data sources to study maternal outcomes and access to care during the prenatal, birth, and postpartum periods in order to identify commonalities among women who experienced SMM and use those findings to create a risk profile of women who are more likely to experience SMM; examine the implementation of maternal safety bundles on SMM and MM outcomes for women up to 1 year postpartum (Intervention 1); gather in-depth data from obstetric care providers on factors that support or hinder safety bundle implementation (Intervention 1); and gather in-depth data from individual women and doulas on facilitators of barriers to the use of doulas to improve care and address inequities (Intervention 2).

DETAILED DESCRIPTION:
Background / Literature Review / Rationale for the study:

Black women experience stark disparities in pregnancy complications and outcomes compared to White women. Recognizing, tracking and understanding patterns of severe maternal morbidity (SMM) and associated inequities by race/ethnicity, along with developing and carrying out interventions to improve the quality of maternal care, are essential to reducing SMM and thereby maternal mortality. To date, there has been little research specifically aimed at understanding whether the maternal health inequities as experienced by Black women can be ameliorated through an integrated care model that includes engagement of providers in the planning and implementation of maternal safety bundles or engaging mothers in prenatal, birth and postpartum support from community doulas. The investigators will use the Health Impact Pyramid and CFIR Framework (Consolidated Framework for Implementation) to develop, implement and assess the effectiveness of such a system in reducing disparities in SMM and mortality. The data sources for this study will include state-level and hospital-specific discharge data collected as part of the Alliance for Innovation on Maternal Health (AIM) project and the Pregnancy to Early Life Longitudinal (PELL) data system, which focuses on population-level data needed to examine health inequities among racial and ethnic minorities in Massachusetts. In addition to these existing data sources, the investigators intend to establish a data collection tool to assess doula services as well as analyze qualitative data from interviews with Black women, and focus groups with obstetrical care providers and doulas to explore the effect of implementing safety bundles and incorporating doula-provided services into prenatal, birth and postpartum care.

ELIGIBILITY:
Intervention I (Maternal Safety Bundles) AIM Bundle Structure, Process and SMM 21 Outcome Measures • Inclusion criteria: Births at the five participating hospital sites for Intervention 1, collecting data one year prior to, during and one year after the study period.

PREM PROM (Patient Reported Experience Measure ( PREM) Patient Reported Outcome Measure (PROM) Surveys for Intervention I

• Inclusion criteria for Pre- and post- surveys for Maternal Safety Bundles Implementation: Birthing individuals who have delivered six weeks to one year prior to the interview at the five participating sites in Intervention 1

Focus groups for Intervention I

• Inclusion criteria: Obstetrical care providers including nurses, midwives, family practitioners, attending obstetricians and trainee obstetricians employed at the five participating hospital sites will be invited to participate in focus groups.

Intervention II (Community doula support) Severe Maternal Mortality (SMM) 21 Outcome Measures • Inclusion criteria: Live births among birthing individuals who identify as Black or African American and who are offered community doula-support at one of the participating four hospitals, either through a hospital-based program or a payer navigation program. The study will include in the intervention arm 340 pregnant women who (1) live in the state of MA, (2) identify as Black or African American, (3) are offered doula care by either their provider or their payer-based navigation program and (4) deliver at one of the four delivering hospitals (Beth Israel Lahey, Boston Medical Center, St. Elizabeth's Medical Center, and Baystate Medical Center). Concurrently, the 340 birthing individuals who were offered doula care in the intervention arm will be matched with birthing individuals who identify as Black or African American, have a live birth, and deliver at one of four hospitals and have similar demographics such as age, comorbidities, payer status, etc.

Focus groups for Intervention II • Inclusion criteria: Persons who practice or identify as community doulas and work with clients who deliver in the state of Massachusetts and have assisted a client in pregnancy, birth, or postpartum within the past 12 months prior to the focus group discussion; obstetrical care provider including nurses, midwives, family medicine practitioners, attending obstetricians, and obstetricians employed at the four participating hospital sites as well as community doula programmatic staff who are employed at participating hospitals sites, or participating community doula organizations, or payers

PREM PROM (Patient Reported Experience Measure Patient Reported Outcome Measure) Surveys for Intervention II

• Inclusion criteria: Live births among birthing individuals who identify as Black or African American and who are offered community doula-support at one of the participating four hospitals, either through a hospital-based program or a payer navigation program.

Intervention I (Maternal Safety Bundles) AIM Bundle Structure, Process and SMM 21 Outcome Measures

• Exclusion criteria: Pregnancies ending prior to 20 weeks and due to ectopic pregnancy not occurring on labor and delivery units of the five participating hospitals

PREM PROM (Patient Reported Experience Measure Patient Reported Outcome Measure) Surveys for Intervention I

• Exclusion criteria: Pregnancies ending prior to 20 weeks and due to ectopic pregnancy not occurring on labor and delivery units of the five participating hospitals

Focus groups for Intervention I

• Exclusion criteria: Staff who have contact with patients but do not identify in the provider types listed in the inclusion criteria

Intervention II (Community doula support) SMM 21 Outcome Measures • Exclusion criteria: Pregnancies ending prior to 20 weeks and due to ectopic pregnancy not occurring on labor and delivery units of the five participating hospitals

Focus groups for Intervention II • Exclusion criteria: Staff who have contact with clients but do not identify in the provider types listed in the inclusion criteria

PREM PROM (Patient Reported Experience Measure Patient Reported Outcome Measure) Surveys for Intervention II

• Exclusion criteria: Pregnancies ending prior to 20 weeks and due to ectopic pregnancy not occurring on labor and delivery units of the four participating hospitals

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1538 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient experience - Respect | 6 -12 weeks postpartum
  Measure through the mothers on respect index (MORi). Range is 14-84 with higher scores indicating more respect.
Patient experience - Autonomy | 6 -12 weeks postpartum
  Mothers autonomy in decision making (MADM). The range is 7- 42 with higher score indicating more opportunities to take an active role and lead decisions.
Severe maternal morbidity (SMM) 20 | At delivery
  Severe maternal morbidity (SMM) includes unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health. Based on 20 ICD 10 codes as defined by the CDC.
Cesarean Birth | At delivery
  The proportion of women with live births who have a C-section.
Severe maternal morbidity (SMM) 21 | At delivery
  Severe maternal morbidity (SMM) includes unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health. Based on 21 ICD 10 codes as defined by the CDC.

SECONDARY OUTCOMES:
Nulliparous, Term, Singleton, Vertex (NTSV) Cesarean Birth Rate | At delivery
  Of all NTSV births the proportion that result in C-section
Severe Maternal Morbidity among Hemorrhage Cases | Monthly up to 6 months
  Denominator: All mothers during their birth admission, excluding ectopics and miscarriages, meeting one of the following criteria:
  * Presence of an Abruption, Previa or Antepartum hemorrhage diagnosis code
  * Presence of transfusion procedure code without a sickle cell crisis diagnosis code
  * Presence of a Postpartum hemorrhage diagnosis code Numerator: Among the denominator, all cases with any SMM code
Severe Maternal Morbidity (excluding cases with only a transfusion code) among Hemorrhage Cases. | Monthly up to 6 months
  Denominator: All mothers during their birth admission, excluding ectopics and miscarriages, meeting one of the following criteria:
  * Presence of an Abruption, Previa or Antepartum hemorrhage diagnosis code
  * Presence of transfusion procedure code without a sickle cell crisis diagnosis code
  * Presence of a Postpartum hemorrhage diagnosis code Numerator: Among the denominator, all cases with any non-transfusion SMM code
Process Measure for Obstetric Hemorrhage - Unit Drills | Monthly up to 6 months
  Report number of Drills and the drill topics P1a: In this quarter, how many OB drills (In Situ and/or Sim Lab) were performed on your unit for any maternal safety topic? P1b: In this quarter, what topics were covered in the OB drills?
Process Measure for Obstetric Hemorrhage - Provider Education | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) At the end of this reporting period, what cumulative proportion of delivering physicians and midwives has completed within the last 2 years an education program on Obstetric Hemorrhage that includes the unit-standard protocols and measures?
Process Measure for Obstetric Hemorrhage - Nursing Education | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) At the end of this reporting period, what cumulative proportion of OB nurses (including L&D and Postpartum) has completed within the last 2 years an education program on Obstetric Hemorrhage that includes the unit-standard protocols and measures?
Process Measure for Obstetric Hemorrhage - Risk Assessment | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) At the end of this quarter, what cumulative proportion of mothers had a hemorrhage risk assessment with risk level assigned, performed at least once between admission and birth and shared among the team?
Process Measure for Obstetric Hemorrhage - Quantified Blood Loss Measurement Utilization | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) In this quarter, what proportion of mothers had measurement of blood loss from birth through the recovery period using quantitative and cumulative techniques?
Structure Measure for Obstetric Hemorrhage - Patient, Family & Staff Support System | Monthly up to 6 months
  Report Completion Date Has your hospital developed OB specific resources and protocols to support patients, family and staff through major OB complications?
Structure Measure for Obstetric Hemorrhage - Debriefs System | Monthly up to 6 months
  Report Start Date Has your hospital established a system in your hospital to perform regular formal debriefs after cases with major complications?
Structure Measure for Obstetric Hemorrhage - Multidisciplinary Case Reviews | Monthly up to 6 months
  Report Start Date Has your hospital established a process to perform multidisciplinary systems-level reviews on cases of severe maternal morbidity (including, at a minimum, birthing patients admitted to the ICU or receiving ≥ 4 units RBC transfusions?
Structure Measure for Obstetric Hemorrhage - Hemorrhage Cart | Monthly up to 6 months
  Report Completion Date Does your hospital have OB hemorrhage supplies readily available, typically in a cart or mobile box?
Structure Measure for Obstetric Hemorrhage - Unit Policy and Procedure | Monthly up to 6 months
  Report Completion Date Does your hospital have an OB hemorrhage policy and procedure (reviewed and updated in the last 2-3 years) that provides a unit-standard approach using a stage-based management plan with checklists?
Structure Measure for Obstetric Hemorrhage - EHR Integration | Monthly up to 6 months
  Report Completion Date Were some of the recommended OB Hemorrhage bundle processes (i.e. order sets, tracking tools) integrated into your hospital's Electronic Health Record system?
Outcome Measure for Severe Hypertension/Preeclampsia - Severe Maternal Morbidity (excluding transfusion codes) among Preeclampsia Cases | Monthly up to 6 months
  Denominator: All mothers during their birth admission, excluding ectopics and miscarriages, with one of the following diagnosis codes:
  * Severe Preeclampsia
  * Eclampsia
  * Preeclampsia superimposed on pre-existing hypertension Numerator: Among the denominator, all cases with any non-transfusion SMM code
Outcome Measure for Severe Hypertension/Preeclampsia - Severe Maternal Morbidity among Preeclampsia Cases | Monthly up to 6 months
  Denominator: All mothers during their birth admission, excluding ectopics and miscarriages, with one of the following diagnosis codes:
  * Severe Preeclampsia
  * Eclampsia
  * Preeclampsia superimposed on pre-existing hypertension Numerator: Among the denominator, all cases with any non-transfusion SMM code
Process Measure for Severe Hypertension/Preeclampsia - Treatment of Severe HTN | Monthly up to 6 months
  Report N/D Denominator: Birthing patients with acute-onset severe hypertension that persists for 15 minutes or more, including those with preeclampsia, gestational or chronic hypertension Numerator: Among the denominator, birthing patients who were treated within 1 hour with IV Labetalol, IV Hydralazine, or PO Nifedipine. The 1 hour is measured from the first severe range BP reading, assuming confirmation of persistent elevation through a second reading.
SMM 20 by Race and Ethnicity | Monthly up to 2 years
  Severe maternal morbidity (SMM) by Race and Ethnicity includes unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health. Based on 20 ICD 10 codes as defined by the CDC.
SMM 21 by Race and Ethnicity | Monthly up to 2 years
  Severe maternal morbidity (SMM) by Race and Ethnicity includes unexpected outcomes of labor and delivery that result in significant short- or long-term consequences to a woman's health. Based on 21 ICD 10 codes as defined by the CDC.
Process Measure for Severe Hypertension/Preeclampsia - Unit Drills | Monthly up to 6 months
  Report number of Drills and the drill topics P1a: In this quarter, how many OB drills (In Situ and/or Sim Lab) were performed on your unit for any maternal safety topic? P1b: In this quarter, what topics were covered in the OB drills?
Process Measure for Severe Hypertension/Preeclampsia - Provider Education | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) At the end of this reporting period, what cumulative proportion of delivering physicians and midwives has completed within the last two years an education program on Severe Hypertension/Preeclampsia that includes the unit-standard protocols and measures?
Process Measure for Severe Hypertension/Preeclampsia - Nursing Education | Monthly up to 6 months
  Report estimate in 10 percent increments (round up) At the end of this reporting period, what cumulative proportion of OB nurses (including L&D and postpartum) has completed within the last two years an education program on Severe Hypertension/Preeclampsia that includes the unit-standard protocols and measures?

CONTACTS AND LOCATIONS:
Overall Officials: Ndidiamaka Amutah Onukagha, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandes KG, Sousa MH, Cecatti JG. Skin Color and Maternal Near Miss: Exploring a Demographic and Health Survey in Brazil. Rev Bras Ginecol Obstet. 2017 May;39(5):209-216. doi: 10.1055/s-0037-1603498. Epub 2017 May 22. PMID 28561138
- [Background] Thomas MP, Ammann G, Brazier E, Noyes P, Maybank A. Doula Services Within a Healthy Start Program: Increasing Access for an Underserved Population. Matern Child Health J. 2017 Dec;21(Suppl 1):59-64. doi: 10.1007/s10995-017-2402-0. PMID 29198051
- [Background] Burns JJ, Livingston R, Amin R. The Proximity of Spatial Clusters of Low Birth Weight and Risk Factors: Defining a Neighborhood for Focused Interventions. Matern Child Health J. 2020 Aug;24(8):1065-1072. doi: 10.1007/s10995-020-02946-y. PMID 32350727
- [Background] Elkafrawi D, Sisti G, Araji S, Khoury A, Miller J, Rodriguez Echevarria B. Risk Factors for Neonatal/Maternal Morbidity and Mortality in African American Women with Placental Abruption. Medicina (Kaunas). 2020 Apr 13;56(4):174. doi: 10.3390/medicina56040174. PMID 32295061
- [Background] Ferranti EP, Frediani JK, Mitchell R, Fernandes J, Li S, Jones DP, Corwin E, Dunlop AL. Early Pregnancy Serum Metabolite Profiles Associated with Hypertensive Disorders of Pregnancy in African American Women: A Pilot Study. J Pregnancy. 2020 Feb 19;2020:1515321. doi: 10.1155/2020/1515321. eCollection 2020. PMID 32148965
- [Background] Gyamfi-Bannerman C, Srinivas SK, Wright JD, Goffman D, Siddiq Z, D'Alton ME, Friedman AM. Postpartum hemorrhage outcomes and race. Am J Obstet Gynecol. 2018 Aug;219(2):185.e1-185.e10. doi: 10.1016/j.ajog.2018.04.052. Epub 2018 May 9. PMID 29752934
- [Background] Wallace ME, Crear-Perry J, Green C, Felker-Kantor E, Theall K. Privilege and deprivation in Detroit: infant mortality and the Index of Concentration at the Extremes. Int J Epidemiol. 2019 Feb 1;48(1):207-216. doi: 10.1093/ije/dyy149. PMID 30052993
- [Background] Ratnasiri AWG, Parry SS, Arief VN, DeLacy IH, Lakshminrusimha S, Halliday LA, DiLibero RJ, Basford KE. Temporal trends, patterns, and predictors of preterm birth in California from 2007 to 2016, based on the obstetric estimate of gestational age. Matern Health Neonatol Perinatol. 2018 Dec 12;4:25. doi: 10.1186/s40748-018-0094-0. eCollection 2018. PMID 30564431
- [Background] Howell EA, Egorova NN, Balbierz A, Zeitlin J, Hebert PL. Site of delivery contribution to black-white severe maternal morbidity disparity. Am J Obstet Gynecol. 2016 Aug;215(2):143-52. doi: 10.1016/j.ajog.2016.05.007. Epub 2016 May 12. PMID 27179441
- [Background] Gillespie SL, Christian LM, Alston AD, Salsberry PJ. Childhood stress and birth timing among African American women: Cortisol as biological mediator. Psychoneuroendocrinology. 2017 Oct;84:32-41. doi: 10.1016/j.psyneuen.2017.06.009. Epub 2017 Jun 15. PMID 28651102
- [Background] Small MJ, James AH, Kershaw T, Thames B, Gunatilake R, Brown H. Near-miss maternal mortality: cardiac dysfunction as the principal cause of obstetric intensive care unit admissions. Obstet Gynecol. 2012 Feb;119(2 Pt 1):250-5. doi: 10.1097/AOG.0b013e31824265c7. PMID 22270275
- [Background] Hans SL, Edwards RC, Zhang Y. Randomized Controlled Trial of Doula-Home-Visiting Services: Impact on Maternal and Infant Health. Matern Child Health J. 2018 Oct;22(Suppl 1):105-113. doi: 10.1007/s10995-018-2537-7. PMID 29855838
- [Background] Poon LC, Kametas NA, Chelemen T, Leal A, Nicolaides KH. Maternal risk factors for hypertensive disorders in pregnancy: a multivariate approach. J Hum Hypertens. 2010 Feb;24(2):104-10. doi: 10.1038/jhh.2009.45. Epub 2009 Jun 11. PMID 19516271
- [Background] Mehta PK, Kieltyka L, Bachhuber MA, Smiles D, Wallace M, Zapata A, Gee RE. Racial Inequities in Preventable Pregnancy-Related Deaths in Louisiana, 2011-2016. Obstet Gynecol. 2020 Feb;135(2):276-283. doi: 10.1097/AOG.0000000000003591. PMID 31923055
- [Background] Bernet P, Gumus G, Vishwasrao S. Maternal Mortality and Public Health Programs: Evidence from Florida. Milbank Q. 2020 Mar;98(1):150-171. doi: 10.1111/1468-0009.12442. Epub 2020 Jan 14. PMID 31943403
- [Background] Murthy NC, Black C, Kahn KE, Ding H, Ball S, Fink RV, Devlin R, D'Angelo D, Fiebelkorn AP. Tetanus, Diphtheria, and Acellular Pertussis and Influenza Vaccinations among Women With a Live Birth, Internet Panel Survey, 2017-2018. Infect Dis (Auckl). 2020 Feb 10;13:1178633720904099. doi: 10.1177/1178633720904099. eCollection 2020. PMID 32095076
- [Background] Murugappan G, Li S, Lathi RB, Baker VL, Luke B, Eisenberg ML. Increased risk of severe maternal morbidity among infertile women: analysis of US claims data. Am J Obstet Gynecol. 2020 Sep;223(3):404.e1-404.e20. doi: 10.1016/j.ajog.2020.02.027. Epub 2020 Feb 27. PMID 32112734
- [Background] Howell EA, Janevic T, Blum J, Zeitlin J, Egorova NN, Balbierz A, Hebert PL. Double Disadvantage in Delivery Hospital for Black and Hispanic Women and High-Risk Infants. Matern Child Health J. 2020 Jun;24(6):687-693. doi: 10.1007/s10995-020-02911-9. PMID 32303940
- [Background] Lyons AB, Peacock A, McKenzie SA, Jacobsen G, Naik HB, Shi VY, Hamzavi IH, Hsiao JL. Evaluation of Hidradenitis Suppurativa Disease Course During Pregnancy and Postpartum. JAMA Dermatol. 2020 Jun 1;156(6):681-685. doi: 10.1001/jamadermatol.2020.0777. PMID 32347884
- [Background] Feinstein L, McWhorter KL, Gaston SA, Troxel WM, Sharkey KM, Jackson CL. Racial/ethnic disparities in sleep duration and sleep disturbances among pregnant and non-pregnant women in the United States. J Sleep Res. 2020 Oct;29(5):e13000. doi: 10.1111/jsr.13000. Epub 2020 Feb 29. PMID 32112620
- [Background] Cesar JA, Camerini AV, Paulitsch RG, Terlan RJ. Non-performance of serological tests for syphilis during prenatal care: prevalence and associated factors. Rev Bras Epidemiol. 2020 Feb 21;23:e200012. doi: 10.1590/1980-549720200012. eCollection 2020. English, Portuguese. PMID 32130400
- [Background] Daw JR, Kolenic GE, Dalton VK, Zivin K, Winkelman T, Kozhimannil KB, Admon LK. Racial and Ethnic Disparities in Perinatal Insurance Coverage. Obstet Gynecol. 2020 Apr;135(4):917-924. doi: 10.1097/AOG.0000000000003728. PMID 32168215
- [Background] Zhou X, McQueen DB, Schufreider A, Lee SM, Uhler ML, Feinberg EC. Black recipients of oocyte donation experience lower live birth rates compared with White recipients. Reprod Biomed Online. 2020 May;40(5):668-673. doi: 10.1016/j.rbmo.2020.01.008. Epub 2020 Jan 23. PMID 32278673
- [Background] Meeks JR, Bambhroliya AB, Alex KM, Sheth SA, Savitz SI, Miller EC, McCullough LD, Vahidy FS. Association of Primary Intracerebral Hemorrhage With Pregnancy and the Postpartum Period. JAMA Netw Open. 2020 Apr 1;3(4):e202769. doi: 10.1001/jamanetworkopen.2020.2769. PMID 32286658
- [Background] Lundeen EA, Park S, Woo Baidal JA, Sharma AJ, Blanck HM. Sugar-Sweetened Beverage Intake Among Pregnant and Non-pregnant Women of Reproductive Age. Matern Child Health J. 2020 Jun;24(6):709-717. doi: 10.1007/s10995-020-02918-2. PMID 32303941